CLINICAL TRIAL: NCT04576936
Title: AIRVO Device Intervention for Moderate to Severe COPD - Pilot Study
Brief Title: AIRVO Device Intervention for Moderate to Severe COPD
Acronym: AIRVO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Renown Health (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1659381-1
Record Dates: First submitted 2020-09-17; First posted 2020-10-06 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: COPD; COPD Exacerbation
Keywords: AIRVO
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AIRVO Device (Experimental): All participants are assigned to this single-arm: Enrolled participants will be given a MyAIRVO2 Device and device stand, and asked to use their device daily, for 12 months
  Interventions: Other: AIRVO

INTERVENTIONS:
Other: AIRVO — Daily, at-home device use of AIRVO device in moderate to severe COPD patients.

SUMMARY:
This is an open (non-blinded), single-arm, clinical trial to assess the efficacy of daily use of a high-flow nasal cannula (HFNC) device in patients with moderate to severe COPD, in addition to standard care, in reducing the amount of COPD exacerbations over a one-year period. Once enrolled in the study, all subjects will be asked to undergo a baseline walking test to measure pulmonary function (6MWT), verify their personal and medical history (demographics), as well as fill in some questionnaires regarding their COPD and its symptoms (SGRQ-C, CAT). All subjects will then receive their own AIRVO2 device, as well as training and instructions on how to use the device at home. Subjects will use the MyAIRVO2 device daily for the following 12 months. Follow-up visits will occur five times over the 12-month study period and will be similar to the baseline visit. Additional data will be collected by the study team for each subject from their electronic medical record during the 12-month study enrollment period. Only information regarding COPD-related medical and/or pharmacy costs, specifically to measure the amount of COPD exacerbations experienced by each subject, will be reviewed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* • Moderate to severe COPD

  * ≥2 inpatient or outpatient claims (ER, or urgent care included) in the previous calendar year
  * ≥2 COPD exacerbations in previous year
  * Current established care within the Reno/Sparks area
  * Residing in Washoe County or Carson City County
  * Ability to travel to site
  * Willing to use myAirVo™2 for at least four hours per day but preferably ≥7 hours or overnight and be capable of handling the myAirVo™2 device after instruction
  * Prior PFT data available prior to admission into project
  * Understand and accept oral and written information in English
  * Life expectancy greater than 1 year

Exclusion Criteria:

* • End-stage renal disease (ESRD)

  * Comorbidity (known malignant disease, terminal illness, dementia, uncontrolled mental illness, COVID-19)
  * Oxygen requirements greater than 6 L/min
  * Bipap or CPAP use in home
  * Receiving hospice care
  * PCP/PI determines the patient is not a good candidate for project inclusion
  * Lung CA
  * Active smoker status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Efficacy of reducing COPD exacerbations as assessed by quantity of exacerbations seen in electronic medical record | 2 years
  evaluate the efficacy of this device on reducing the number of COPD exacerbations, and/or COPD-related emergency department (ED) visits and hospitalizations, over a 12-month period compared with the previous 12 months

SECONDARY OUTCOMES:
COPD Health-related Quality of Life | 1 year
  evaluate whether the use of myAirvo™2 may improve health-related quality of life (HRQoL) in COPD patients based on responses to the St. George's Respiratory Questionnaire - COPD (SGRQ-C). Higher scores on this measure indicate greater impairment.
COPD Health-related Quality of Life | 1 year
  evaluate whether the use of myAirvo™2 may improve health-related quality of life (HRQoL) in COPD patients based on responses to the COPD Assessment Test (CAT). Higher scores on this measure indicate greater impairment.
Respiratory function test results | 1 year
  evaluate the efficacy of daily myAirvo™2 use on respiratory function using the Six Minute Walk Test

CONTACTS AND LOCATIONS:
Locations (1):
- Renown Medical Group - Pulmonary & Sleep Medicine, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No